CLINICAL TRIAL: NCT06159153
Title: Dynamic Ultrasonography VS MRI in the Evaluation of Meniscal Lesions in Patients With an Indication for Arthroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: US- DYNAMIC
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Meniscus Lesion; Meniscus Disorder; ACL Injuries
Keywords: dynamic ultrasonography; arthroscopy; MRI; Interventional trial
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dynamic Ultrasonography assessment (Experimental): Patients admitted for ACL injury and indication for arthroscopy will have dynamic ultrasound evaluation that will be compared with an MRI.
  Interventions: Diagnostic Test: Dynamic Ultrasonography assessment

INTERVENTIONS:
Diagnostic Test: Dynamic Ultrasonography assessment — Ultrasound evaluation that will be compared with an MRI.

SUMMARY:
This is a diagnostic, open-label, single-center interventional study.

This study aims to evaluate the diagnostic accuracy of dynamic ultrasonography for meniscal injuries in patients with an indication for arthroscopy, and to compare it with the study in MRI.

DETAILED DESCRIPTION:
Patients admitted for ACL injury and indication for arthroscopy will be included in a study involving the evaluation of the diagnostic accuracy of dynamic ultrasound compared with MRI.

A total of 254 patients will be included, who after providing their signed informed consent to participate in the study, will undergo dynamic ultrasound. After giving signed consent to participate in the study, the patient will undergo the ultrasound evaluation for assessment of possible meniscal injury; Radiological examinations in the patient's possession or from the patient's medical record will be collected during or before the diagnostic investigation.

ELIGIBILITY:
Inclusion Criteria:

Patients with an indication for knee arthroscopy with:

1. Age between 18 and 60 years;
2. Unilateral involvement;
3. Presence of symptomatology such that dynamic ultrasound examination is precluded;
4. Ability and consent of patients to actively participate in the study;

Exclusion Criteria:

1. Patients unable to express consent;
2. Patients with malignant neoplasms;
3. Patients with rheumatic diseases;
4. Patients with diabetes;
5. Patients with metabolic disorders of the thyroid gland;
6. Patients abusing alcoholic beverages, drugs or medications;
7. Body Mass Index > 35;
8. Pregnant or lactating women;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 254 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity of Dynamic Ultrasonography assessment | baseline
  Baseline ultrasonography evaluation for assessment of possible meniscal injury. The ultrasound examination will be compared with an MRI using the arthroscopy result as the gold standard.
Diagnostic specificity of Dynamic Ultrasonography assessment | baseline
  Baseline ultrasonography evaluation for assessment of possible meniscal injury. The ultrasound examination will be compared with an MRI using the arthroscopy result as the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Andriolo, MD, Principal Investigator — Istituto Ortopedico Rizzoli - II Clinica Ortopedica e Traumatologica
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dong F, Zhang L, Wang S, Dong D, Xu J, Wu H, Liu Y, Li M. The diagnostic accuracy of B-mode ultrasound in detecting meniscal tears: a systematic review and pooled meta-analysis. Med Ultrason. 2018 May 2;20(2):164-169. doi: 10.11152/mu-1252. PMID 29730682
- [Background] Cook JL, Cook CR, Stannard JP, Vaughn G, Wilson N, Roller BL, Stoker AM, Jayabalan P, Hdeib M, Kuroki K. MRI versus ultrasonography to assess meniscal abnormalities in acute knees. J Knee Surg. 2014 Aug;27(4):319-24. doi: 10.1055/s-0034-1367731. Epub 2014 Jan 28. PMID 24474166
- [Background] Sharifah MI, Lee CL, Suraya A, Johan A, Syed AF, Tan SP. Accuracy of MRI in the diagnosis of meniscal tears in patients with chronic ACL tears. Knee Surg Sports Traumatol Arthrosc. 2015 Mar;23(3):826-30. doi: 10.1007/s00167-013-2766-7. Epub 2013 Nov 17. PMID 24240983
- [Background] Schroeder A, Musahl V, Urbanek C, Onishi K. Dynamic Sonographic Visualization of an Occult Posterior Lateral Meniscocapsular Separation: A Case Report. PM R. 2018 Nov;10(11):1288-1291. doi: 10.1016/j.pmrj.2018.03.017. Epub 2018 Apr 5. PMID 29626617
- [Background] Alizadeh A, Babaei Jandaghi A, Keshavarz Zirak A, Karimi A, Mardani-Kivi M, Rajabzadeh A. Knee sonography as a diagnostic test for medial meniscal tears in young patients. Eur J Orthop Surg Traumatol. 2013 Dec;23(8):927-31. doi: 10.1007/s00590-012-1111-z. Epub 2012 Oct 27. PMID 23412237
- [Background] Wareluk P, Szopinski KT. Value of modern sonography in the assessment of meniscal lesions. Eur J Radiol. 2012 Sep;81(9):2366-9. doi: 10.1016/j.ejrad.2011.09.013. Epub 2011 Oct 5. PMID 21982460